CLINICAL TRIAL: NCT06437431
Title: Glenzocimab in Anterior Stroke With Large Ischemic Core Eligible for Endovascular Therapy
Acronym: GALICE
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JDS_2023_13
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — glenzocimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- glenzocimab (Experimental)
  Interventions: Drug: glenzocimab
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: glenzocimab — Two vials (2x500 mg) of glenzocimab should be administered concomitantly for eligible patients for a total dose of 1g of glenzocimab as an IV infusion over 6 hours, with 1/4 of the dose administered by a 15-minutes bolus and 3/4 of the dose administered by 5h45minutes continuous infusion.
  Arms: glenzocimab
Drug: placebo — Placebo of glenzocimab is 0.9% NaCl for IV administration. It is supplied for clinical trial use in vials of 50 mL. Two vials of placebo should be administered concomitantly for eligible patients. The administration scheme will be the same as in the experimental arm.
  Arms: placebo

SUMMARY:
Until recently, acute ischemic stroke (AIS) patients with a baseline large infarct core have been generally excluded from clinical trials of endovascular therapy (EVT). A first multicenter randomized trial (Rescue Japan Limit trial) found a significant benefit of EVT in AIS patients with large infarct core (DWI-ASPECTS of 3-5). Another non-randomized multicenter prospective study found a positive association of EVT with 3-month outcome in AIS patients with a baseline CTP ischemic core volume >70mL. More recently, 2 additional randomized trials were published. They both confirmed a strong efficacy of EVT in patients with large infarct core. However, even with EVT, the proportion of good outcome (3-month mRS score of 0-3), remains low in these highly severe AIS patients ranging from 8-30%. Almost 75% of EVT-treated patients are still severely disabled or dead at 3 months. In experimental studies, we and others described the pathophysiological features of the downstream microvascular thrombosis (DMT) in AIS setting highlighting its immediate occurrence and the pivotal role of platelet activation and aggregation. In recent clinical studies, it has been shown that, even with a complete angiographic recanalization after EVT, up to 40% of patients presented no-reflow (NR), a failure of downstream microvascular reperfusion, visible on perfusion imaging performed after EVT. Some clinical studies reported the clinical impact of NR after successful EVT. We found that DMT participated to the development of neurovascular lesions in AIS with both an early ischemic lesion growth risk evolving towards a delayed hemorrhagic transformation (HT) and vasogenic edema risks and therefore worse outcome. Our results suggested that an antiplatelet therapy infused early in AIS patients could reduce both the ischemic lesion but also the risk of delayed vasogenic edema and HT. Platelet glycoprotein VI (GPVI) is a key receptor for collagen and fibrin and plays a major role in platelet activation, platelet recruitment and thrombosis. Furthermore, inhibition of the GPVI does not impair haemostasis and subjects with a genetic or acquired GPVI deficiency are not prone to excessively bleed.

Glenzocimab is a monoclonal antibody directed against the GPVI. It has been developed as an immediate antiplatelet agent with minimal bleeding risk for treating AIS. The ACTIMIS trial, a phase IB/IIA clinical study that assessed for the first time the glenzocimab IV infusion in AIS patients found very promising safety data including a significant reduce of symptomatic HT (1% vs. 7.8%) and mortality rates (7.8% vs. 18.7%), especially in severe AIS patients. Our hypothesis is that IV glenzocimab infusion would improve good functional outcome in large ischemic core AIS patients treated with EVT by reducing the DMT, ischemic lesion growth, and the HT rate.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Acute ischemic stroke due to an isolated proximal anterior large vessel occlusion (M1 and M2 segment of the middle cerebral artery, terminal internal carotid artery (TICA))
* Indication of EVT within the time window of 0 to 24 hours in participants treated with or without intravenous thrombolysis.
* Presenting with a baseline infarct core volume assessed on the MRI (DWI sequence) or CT scan with an ASPECTS<6
* Woman <49 years old must have a negative serum/urine pregnancy test at baseline

Exclusion Criteria:

* Possible tandem occlusion on the baseline imaging, potentially requiring stenting
* Significant pre-stroke disability (mRS>2)
* Patients under or needing immediate dual anti-platelet therapy (DAPT) within the first 24 hours after the cessation of glenzocimab or placebo infusion
* Significant mass effect with midline shift as confirmed on CT/MRI
* Gastrointestinal or urinary tract haemorrhage in previous 21 days
* Patient with intracranial haemorrhage
* Platelet count <100 000 mm3
* Known hypersensitivity to glenzocimab or to any of the excipients
* Known hypersensitivity to the gadolinium used for the brain MRI perfusion, or one of its excipients
* Known Severe renal insufficiency (Grades 4-5) with a glomerular filtration rate < 30mL/Min/1.73m2
* Patients receiving anticoagulants within the last 24 hours and:

  * For heparin, an elevated aPTT -greater than upper limit of normal for laboratory
  * For vitamin K antagonists (ex: warfarin), an INR >1.7;
  * For direct thrombin inhibitors or direct factor Xa inhibitors, a plasmatic dosage of the drug greater than upper limit of normal for laboratory
* Pregnant or breastfeeding woman
* Participation in another interventional clinical investigational drug or medical device trial within 30 days prior to the inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
proportion of good functional outcome at 3 months. | Month 3
  Functional outcome at 3 months will be assessed with the modified Rankin Scale (mRS) score dichotomized 0 to 3 versus 4 to 6, collected by phone by trained certified professionals and blinded to the treatment allocation and centralized.
  In case of loss of follow-up and impossibility to obtain mRS from the patient or his family at three month, a mRS score from the patient medical record (e.g. follow-up neurologist consultation, report of the rehabilitation hospitalization etc…) will be used if it is more or less 1 month from the 3-month protocol follow-up date.

IPD SHARING:
Plan to Share IPD: No